CLINICAL TRIAL: NCT06638905
Title: A Prospective, Open Label Clinical Study Evaluating the Efficacy and Safety of Skincare Serum and Cream for Anti-aging of Facial Skin
Brief Title: Efficacy and Safety of Skincare Serum and Cream for Anti-aging of Facial Skin
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Babor Americas (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Babor-2024
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Facial Wrinkles; Skin Aging
Keywords: Wrinkles; Face Wrinkles; Cosmetic; Crow's Feet

STUDY DESIGN:
Intervention Model Description: Subjects will be treated with a combination therapy of Babor Ultimate ECM Repair Serum and the Babor Cure Cream to their entire face.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Babor Products (Experimental): Enrolled subjects will all receive Babor Ultimate ECM Repair Serum and Babor Cure Cream to be applied to their entire face.
  Interventions: Drug: Babor Ultimate ECM Repair Serum; Drug: Babor Cure Cream

INTERVENTIONS:
Drug: Babor Ultimate ECM Repair Serum — The BABOR® Ultimate ECM Repair Serum contains Biogen plant extract, cotton thistle flower, and wakame extract. Babor products are encouraged to be used simultaneously mornings and/or evenings to reinforce the skin's protective barrier, promote vibrant skin, and restore skin elasticity and firmness.
Drug: Babor Cure Cream — Babor products are encouraged to be used simultaneously mornings and/or evenings to reinforce the skin's protective barrier, promote vibrant skin, and restore skin elasticity and firmness.

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of combination therapy of BABOR® Ultimate ECM Repair Serum and the BABOR® Cure Cream for the improvement of anti-aging through the use of investigator assessments, subject questionnaires/assessments, photography, skin imaging, and reported adverse reactions.

DETAILED DESCRIPTION:
Enrolled subjects will use a skin care regimen cosisting of BABOR® Ultimate ECM Repair Serum, BABOR® Cure Cream gel, mineral sunscreen, and regeneration cleanser and regeneration toner. Subjects satisfying all inclusion and exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory photography using Canfield VISIA imaging and handheld 2D photography. Patients will return for follow-up assessments at Day 30, 60, and 90.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 50 years old (inclusive).
* Subjects must be able and willing to provide written informed consent and photography release.
* At the baseline evaluation, all subjects must exhibit mild to moderate skin aging, as defined below (Appendix A):

  1. Class I-II of Wrinkling on the Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale
  2. Score 1-6 of Degree of Elastosis on the Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale
  3. Mild to Moderate on Redness/Erythema Grading Scale
  4. Mild to Moderate on Dryness/Scaling/Roughness Grading Scale
  5. Mild to Moderate on Luminosity Scale
* Subject must be in good general health with no other skin disease, disease state or physical condition which would impair evaluation of the areas to be treated or which would increase the subject's health risk by study participation.
* Subjects must have a willingness to minimize sun exposure, avoid direct sun exposure on the face, and avoid the use of tanning beds for the entire duration of the study. Must be willing to wear a hat and reapply sunscreen if sun exposure is unavoidable.
* Subjects must be willing and able to understand and comply with the requirements of the study including prolonged sun exposure and apply the products as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.

Exclusion Criteria:

* Subjects who are pregnant, planning pregnancy during the course of the study, or breastfeeding.
* Subjects with an active bacterial, fungal, or viral infection in the treatment area
* Subjects with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* Subjects receiving any topical products containing tretinoins or derivatives, alpha-hydroxy acids, salicylic acid, and vitamins C or E (includes derivatives thereof) on the face within 14 days prior to or during the study period, other than the study products.
* Subjects receiving a chemical peel, any systemic steroids, a non-ablative laser, ablative laser, microfocused ultrasound, light or radio frequency treatment, deep chemical peel, and/or has had a Dermabrasion on their face must have discontinued the drug/treatment and/or had the procedure at least 6 months prior to entering the study.
* Subjects who have had a microdermabrasion (light or medium skin peel) treatment on their face within 30 days prior to and not willing to refrain from use for the duration of the study period.
* Subjects with recently excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study or has used self-tanner within 7 days of study entry.
* Subjects that has previously been treated with a systemic retinoid within the past 3 months (e.g., Accutane®, Roche Dermatologics).
* Subjects with a history of keloids or hypertrophic scars.
* Subjects with known allergies to any of the product ingredients.
* Subjects with a tattoo and/or scar in the treatment area that in the investigators opinion would interfere with study assessments.
* Subjects with history of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis) at the discretion of the investigator.
* Inability to comply with all study protocol restrictions and visits.
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.
* History of non-compliance with clinical research protocols.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-03-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Fitzpatrick- Goldman Classification of Wrinkling and Degree of Elastosis Scale | Screening, Day 60, Day 90
  Circle appropriate class:
  Class one: Mild Fine Wrinkles 1-2-3
  Class two: Moderate Wrinkles 4-5-6
  Class three: Severe Wrinkles 7-8-9
Evaluating Investigator Expert Grading Scales | Screening, Day 30, Day 60, Day 90
  Redness/ Erythema:
  None (Score of 0) No erythema or redness of the treatment area Mild (Score of 1, 2 or 3) Slight, but definite redness of the treatment area Moderate (Score of 4, 5 or 6) Definite redness of the treatment area Severe (Score of 7, 8 or 9) Marked redness of the treatment area
  Dryness/ Scaling/Roughness:
  None (Score of 0) No dryness, roughness, or flaking/scaling of the treatment area Mild (Score of 1, 2 or 3) Slight, but definite roughness, some areas of light visible flaking/scaling of the treatment area Moderate (Score of 4, 5 or 6) Definite roughness and areas of visible flaking/scaling of the treatment area Severe (Score of 7, 8 or 9) Marked roughness and areas of visible flaking/scaling of the treatment area
Evaluating Investigator Expert Grading Scales (part 2) | Screening, Day 30, Day 60, Day 90
  Luminosity:
  None (Score of 0) Radiant, luminous or glowing appearance Mild (Score of 1, 2 or 3) Some areas of dullness or matte skin in the treatment area Moderate (Score of 4, 5 or 6) Several areas of dullness or matte skin in the treatment area Severe (Score of 7, 8 or 9) Dull/matte and/or sallow skin appearance

SECONDARY OUTCOMES:
Evaluating Investigator Tolerability Assessment | Screening, Day 30, Day 60, Day 90
  Stinging/ Burning:
  None (Score of 0) No stinging/burning of the treatment area Mild (Score of 1, 2 or 3) Slight, but definite stinging/burning of the treatment area Moderate (Score of 4, 5 or 6) Definite stinging/burning of the treatment area Severe (Score of 7, 8 or 9) Marked stinging/burning of the treatment area
  Itching:
  None (Score of 0) No itching of the treatment area. Mild (Score of 1, 2 or 3) Slight, but definite itching of the treatment area. Moderate (Score of 4, 5 or 6) Definite itching of the treatment area that is distracting from daily activities.
  Severe (Score of 7, 8 or 9) Marked itching of the treatment area that wakes you up at night.
  Rash:
  None (Score of 0) No new rash over the treatment area. Mild (Score of 1, 2 or 3) New rash covering some of the treatment area. Moderate (Score of 4, 5 or 6) New rash covering much of the treatment area. Severe (Score of 7, 8 or 9) New rash covering the entirety of the treatment area.
Subject Self-Assessment Questionnaire (part 1) | Screening, Day 30, Day 60, Day 90
  1. Skincare regimen helps reduce the wrinkles of my facial skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  2. Skincare regimen helps reduce the dryness of my facial skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  3. Cleanser/moisturizer regimen helps decrease the dullness of my facial skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  4. Skincare regimen helps reduce the unevenness of my facial skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
  5. Skincare regimen leaves my facial skin radiant/brighter. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
Subject Self-Assessment Questionnaire (part 2) | Screening, Day 30, Day 60, Day 90
  6. Skincare regimen leaves my facial skin softer. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 7. Skincare regimen leaves my facial skin smoother. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 8. Skincare regimen is gentle. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 9. Skincare regimen leaves my facial skin healthy looking. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 10. Skincare regimen helps reduce the flakiness of my skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
Subject Self-Assessment Questionnaire (part 3) | Screening, Day 30, Day 60, Day 90
  11. I now understand the importance of a consistent skincare routine. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 12. I feel more confident about the appearance of my facial skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 13. Using this skincare regimen makes me optimistic about my appearance. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 14. This skincare regimen was easy to follow. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 15. It was easy to adhere to this skincare routine. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly
Subject Self-Assessment Questionnaire (part 4) | Screening, Day 30, Day 60, Day 90
  16. Using these products did not irritate my skin. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 17. The results I received made me want to continue this skincare routine. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 18. I was able to easily commit to this routine due to its simplicity. Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly 19. Please include further comments regarding your experience with these products.
  Agree Strongly Agree Neither agree nor disagree Disagree Disagree Strongly

IPD SHARING:
Plan to Share IPD: No